CLINICAL TRIAL: NCT06109922
Title: Investigating the Effects of Dietary Phospholipids on Stress Reactivity and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Volac International Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 66CH2
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Mood; Stress; Physiological Stress
Keywords: mood; stress; stress reactivity; stress recovery; perceived task demand
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, parallel groups design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment will be blinded according to the randomisation schedule by a researcher who has no other involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Bioactive whey protein concentrate containing phospholipids.
  40g pre weighed powder to be mixed with 350ml of water. Consumed once daily for 12 weeks alongside their fattiest meal of the day.
  Interventions: Dietary Supplement: Active
- Placebo (Placebo Comparator): Placebo
  Placebo powder matched for macronutrient and caloric content containing pea protein around 40g powder mixed with 350ml water consumed once daily for 12 weeks alongside fattiest meal of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — 40g bio-active whey protein concentrate powder containing phospholipids
  Other Names: Active Treatment
  Arms: Experimental
Dietary Supplement: Placebo — Around 40g pea protein powder not containing phospholipids
  Other Names: Placebo Treatment
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the effects of 6- and 12- week supplementation of a bioactive whey protein concentrate drink containing dairy phospholipids on stress reactivity and recovery in healthy adults.

The proposed randomised, double-blind, placebo-controlled parallel groups design methodology will assess the stress reactivity and recovery effects (both self-reported and physiological) of 40g per day of bioactive whey protein concentrate in the form of a powder that the participant will be required to mix with 350ml of water and matched placebo prior to (baseline) and after -6 week and -12 week supplementation. The trial will utilise the Multi-tasking framework (MTF) during testing visits to elicit an acute stress response within the laboratory. Self reported anxiety (STAI short-form) at multiple time points before and after the stressor will be measured as well as perceived task demand following the stressor (NASA-TLX).

Physiological measurements of the stress response will also be measured through blood pressure, heart rate arability, and galvanic skin response.

150 participants will participate, aged 25-49, and self-reported as being in good health. Participants will be supplied with either the active treatment or the placebo (allocated by a randomised schedule) whilst visiting the research centre for the testing appointments, and will take treatment home to consume daily for the duration of the study. Participants will record time of taking treatment each day in a treatment diary which will be returned to the research centre, along with any unused treatment, upon completion of the study.

DETAILED DESCRIPTION:
The study will follow a randomised, placebo-controlled, double-blind, parallel groups design. Participants will be given 12-weeks' worth of either placebo or active treatment to be consumed at home each day (double blinded), will attend all 5 appointments required, will complete the at home treatment diary daily, as well as participate in the multi-tasking stress tasks on each of the 3 testing visits.

Participants will attend the research centre on four separate occasions, which will include a screening/training visit, pre intervention testing visit, a mid-point testing visit (at 6 weeks), and a completion of intervention testing visit (at 12 weeks). 5 Appointments in total including the online appointment to check for eligibility. The remote screening session will be completed via telephone call and will comprise briefing on the requirements for the study, answering any initial questions, obtaining of informed consent via completion of an online consent form, health screening, collection of demographic information, and completion of the Caffeine Consumption Questionnaire (CCQ).

The introductory/training visit to the laboratory will begin with physiological eligibility measures that cannot be completed remotely (e.g., blood pressure, height and weight, waist-to-hip ratio) followed by training on the cognitive and mood measures.

The study will include 150 healthy participants aged between 25-49 years, who will receive 12 weeks' worth of either 40g per day of bioactive whey protein concentrate powder containing dairy phospholipids (to be mixed with 350ml of water to form a drink), or a similar of placebo powder. Participants will be randomly allocated to either the treatment or placebo group and neither the participant nor the researcher will know which group they have been allocated to. Full instructions of how and when to take treatment each day will be explained to the participants when treatment is given at testing visit 1.

On each of the three study days (Day 1, 42, and 84) participants will attend the research centre, having abstained from alcohol for 24 hours, and caffeine overnight, following a standardised breakfast of cereal and/or toast at home no later than 1 hour prior to arrival. After completing the cognition tasks outlined in a separate protocol, the participants will be taken one by one to a separate room, accompanied by the lead researcher, to participate in the stress reactivity and recovery task. The task is the Multi-Tasking Framework (MTF) and will last approx. 20 minutes. During this time, participants will be required to remain concentrated on 4 tasks simultaneously to achieve the highest overall score possible. The tasks are a mixture of difficulty and require different skills such as reaction time, memory, and attention. Whilst the participants are completing the tasks, the researcher will be monitoring their performance and providing feedback and instruction. Blood pressure will be taken before and after the task. Questionnaires to measure state anxiety and perceived task demand will be taken at different time points surrounding the stressor. Participants will also be required to wear a heart rate monitor and sensors on their fingertips to measure heart rate variability and galvanic skin response in response to the stressor.

Participants will additionally complete a treatment guess form at their final visit and will be fully debriefed.

ELIGIBILITY:
Inclusion Criteria:

* Participant must self-assess themselves as being in good health
* Participant must be aged 25 to 49 years at the time of giving consent
* Participants first language is English or are fluent in English

Exclusion Criteria:

* Have any pre-existing medical conditions/illness which will impact taking part in the study. Cases can be looked at case-by-case.
* Are currently taking any prescription medications (NOTE the explicit exceptions to this are contraceptive treatments for female participants, and those taking "as needed" in the treatment of asthma and/or hay fever)
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg). NOTE: that we must measure this in the lab using our blood pressure monitors and can only use our measurements to assess eligibility rather than home or doctors readings
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2.
* Are pregnant, seeking to become pregnant or lactating.
* Have been diagnosed with a neurological condition, or assessed as having a learning/behavioral or neurodevelopmental difference (e.g. dyslexia, autism, ADHD)
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products (if you have recently quit smoking or using replacements you must have stopped using them altogether for a period of 3 months before participating in this study)
* Have excessive caffeine intake (>500 mg per day). Note: This will be calculated at screening but feel free to query this with the researcher prior to attendance
* Have relevant food allergies/ intolerance/ sensitivities
* Have taken antibiotics within the past 4 weeks.
* Have taken dietary supplements e.g., vitamins, omega 3 fish oils etc. in the last 4 weeks . (Note: participation is possible following a 4 week wash out prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised. Please discuss with the researcher if unsure. NOTE: we would never advise stopping supplements prescribed by your doctor e.g. iron, calcium etc, only those out of choice).
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months.
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months, including a medical diagnosis of anxiety or depression.
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Have any sleep disorders or take any sleep medications.
* Have any known active infections.
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption
* Follow an "extreme" diet. i.e., high fat, low sugar, low carb, high protein, paleo etc
* Are planning a major lifestyle change regarding diet or exercise regime in the next 3 months.
* Are unable to meet the minimum requirement scores on the cognitive tasks.
* Experienced an event (professional or personal) that is likely to have impacted your emotional and/or psychological state within the last 8-10 weeks (for example but not restricted to change of professional function, death of a family member, divorce, surgery, accident etc)
* Have an upcoming event (personal or professional) that is likely to affect your emotional, psychological state or hormonal state planned during the next 8-10 weeks, including but not limited to job change, house move, important medical exam etc.

  * Have a current diagnosis of renal impairments or phenylketonuria

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Stress Reactivity and Recovery | Following 6- and 12- week supplementation
  Ratings of anxiety as defined by the State trait anxiety inventory (STAI) short form sub scale

SECONDARY OUTCOMES:
Perceived Task Demand | Following the multi-tasking framework at baseline, 6-weeks, and 12- weeks supplementation.
  Treatment effects on perceived task demand of the multi-tasking framework via the NASA task load index (NASA TLX). Five 7- point scales summed to create a measure of perceived mental workload of the multi-tasking framework.
Galvanic Skin Response- Physiological measure of stress response | During each completion of the multi-tasking framework (baseline, 6 weeks, and 12 weeks).
  treatment effects on physiological stress response via galvanic skin response. Measuring readings of galvanic skin response during each completion of the multi-tasking framework (3) to determine physiological response to the psychological stressor pre, mid and post intervention.
Heart Rate Variability- Physiological measure of stress response | During each completion of the multi-tasking framework (baseline, 6 weeks, 12 weeks).
  treatment effects on physiological stress response via heart rate variability. Measuring readings of heart rate variability, via a chest strap sensor and polar watch, during each completion of the multi-tasking framework (3) to determine physiological response to the psychological stressor pre, mid, and post intervention.
Systolic Blood Pressure- Physiological measure of stress response | During each completion of the multi-tasking framework (baseline, 6 weeks, and 12 weeks).
  Treatment effects on physiological response to stress via systolic blood pressure readings. measuring blood pressure pre and post completion of the multi-tasking framework (3) to determine physiological response to the psychological stressor pre, mid and post intervention.
Multi-tasking Framework Overall Scores | At baseline, 6- weeks, and 12- weeks of intervention.
  treatment effects on overall multi-tasking framework scores following 6-, and 12- weeks Treatment effects on overall multi-tasking framework scores following 6- and 12- weeks of intervention. Participants receive scores upon completion of 20 minutes of the multi-tasking framework. 10 points per correct answer and 10 points deducted for every incorrect or missed response. Scores can range from minus to positive. Scores indicate engagement in the tasks. The higher the score the higher the engagement in the tasks.
Diastolic Blood Pressure- Physiological measure of stress response. | During each completion of the Multi-tasking framework (baseline, 6 weeks, and 12 weeks)
  Treatment effects on physiological response to stress via diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No